CLINICAL TRIAL: NCT05377671
Title: Backward Masking Tasks to Decipher Impaired Input-Output Connections in MS @7T
Acronym: BIO7
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A00174-39; 2021-32 (Other: sponsor reference)
Record Dates: First submitted 2022-05-10; First posted 2022-05-17 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Difference in Regional Brain Activity

STUDY DESIGN:
Intervention Model Description: 40 patients (20 patients with a cognitive deficit at least 2 SD below the norm and 20 patients without cognitive impairment) will be explored by multimodal ultra-high field (7T) MRI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive deficit group (Experimental): All patients will undergo task MRI and standard clinical assessments, including neuropsychological examination. The MRI includes, in addition to structural task sequences, diffusion imaging and resting state fMRI.
  Interventions: Diagnostic Test: IRM multimodale a ultra-haute camp
- Without cognitive group (Experimental): All patients will undergo task MRI and standard clinical assessments, including neuropsychological examination. The MRI includes, in addition to structural task sequences, diffusion imaging and resting state fMRI.
  Interventions: Diagnostic Test: IRM multimodale a ultra-haute camp

INTERVENTIONS:
Diagnostic Test: IRM multimodale a ultra-haute camp — The MRI includes, in addition to structural task sequences, diffusion imaging and resting state fMRI.

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory and neurodegenerative disease of the central nervous system. People with MS frequently suffer from cognitive and visual impairment. Moreover, patients rank cognition and vision as two of the three most valuable bodily functions, in addition to mobility. Here the investigator use the established backward masking paradigm to study structural and functional alteration at the sub-milimeter scale in ultra-high field MRI in order to decipher the different input-output loops associated with the preservation and alteration of cognition in MS.

DETAILED DESCRIPTION:
To identify abnormalities in mesoscale input and output connectivity at structural and functional levels that differ between patients with and without cognitive impairment. To address this objective, the investigator will analyse and compare functional activations in the primary visual cortex and task-associated regions in our previous studies. Secondary objectives: To develop, improve and validate multimodal laminar imaging at ultra-high field strength (7T) in comparison to control subjects available in our database to identify and quantify focal impairment in MS.

This is a cross-sectional study. 40 patients (20 patients with a cognitive deficit at least 2 SD below the norm and 20 patients without cognitive impairment) will be explored by multimodal ultra-high field (7T) MRI. The protocol included task, resting FMRI (functional connectivity), diffusion tensor (structural connectivity) and anatomical sequences (lesions and atrophy). In addition, the investigator will analyse standard clinical assessments including a neuropsychological examination. To understand the mechanisms underlying neurodegeneration and adaptation, it is important to contrast physiological and pathological alterations. In addition to comparing cognitively preserved and cognitively impaired patients, the investigator aim to compare our participants to a representative normative dataset available in our database of healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>= 18 years of age) with MS defined according to the McDonald criteria 2017 (Thompson et al., 2018)
* For the group of patients without cognitive impairment: SDMT or PASAT >=0 (based previous clinical assessments)
* For the group of patients with cognitive impairment: SD SDMT or PASAT <= -1.5 (based based on previous clinical assessments) (Parmenter et al., 2007)
* Person without uncontrolled systemic disease such as cancer, autoimmune disease, liver failure, severe or untreated hypertension, conduction conduction disorder or severe rhythm disorder
* No one with chronic psychiatric illness, severe dementia syndrome demented syndrome.
* No contraindication to MRI examination (claustrophobia, metallic foreign bodies, pacemakers),
* A person with social security coverage,
* Person having read, understood and signed an informed consent after information

Exclusion Criteria:

* Pregnant women
* Other inflammatory demyelinating diseases of the CNS
* Usual contraindications for an MRI examination: claustrophobia, metallic foreign bodies pacemakers, severe renal insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Difference in regional brain activity between patients with and without cognitive impairment measured by the Bold signal | 1 year
  The explorations will be performed on a very high field imager (7T Terra, Siemens, Erlangen) dedicated to the research.

SECONDARY OUTCOMES:
Cognitive performance | 1 year
  The precision corresponding to the % of correct answers.
Morphology | 1 year
  Cortical thickness. Next, the investigator will use Freesurfer (www.surfer.nmr.mgh.harvard.edu) to perform a vertex-wise cross-sectional comparison of cortical thickness between the two groups using a general linear model (GLM) controlling for age and sex. In a second model, the association between cortical thickness and time to conscious treatment will be calculated, also corrected for age and sex in the GLM. The results per vertex were corrected by the false discovery rate (FDR) at a threshold of p < 0.05.
Structural connectivity | 1 year
  The investigator will use the average FA to construct weighted connectivity matrices between 160 nodes (80 cortical regions per hemisphere) based on the Destrieux atlas. "Strength", as a measure of regional structural connectivity, was calculated as the sum of weighted connections within and between each node for each subject.
Functional connectivity | 1 year
  First, the investigator will perform preprocessing of the resting fMRI data, including correction for motion distortion and slice synchronization and cor- gistration with T1 volume and regional parcellation using SPM12. Then, all voxels in each region and time points will be averaged after application of the regression procedure for head motion, cerebrospinal fluid signals, white matter signals, and the overall average signal. After the preprocessing step, the output data acquired from the averaged region time series were used to perform wavelet analysis (frequency band: 0.1 Hz - 0.05 Hz, TR=2.5 s) using the brainwaver package in R. To calculate the raw functional connectivity, the investigator will calculate the absolute Pearson correlations between the time series of the wavelet coefficients of each region. For better comparability of the networks, the top 15% of connections defined the connectivity matrices. The degree of the nodes is the primary evaluation criterion.

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — ASSISTANCE PUBLIQUE HOPITAUX MARSEILLE; Jan-Patrick STELLMANN, Principal Investigator — ASSISTANCE PUBLIQUE HOPITAUX MARSEILLE
Locations (1):
- Assistance Publique Hopitaux Marseille, Marseille, Bouches Du Rhône, France